CLINICAL TRIAL: NCT03199469
Title: ASPIRO: A Phase 1/2/3, Randomized, Open-Label, Ascending-Dose, Delayed-Treatment Concurrent Control Clinical Study to Evaluate the Safety and Efficacy of AT132, an AAV8-Delivered Gene Therapy in X-Linked Myotubular Myopathy (XLMTM) Patients
Brief Title: A Study of AT132 in Young Children With X-Linked Myotubular Myopathy (XLMTM)
Acronym: ASPIRO
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Astellas Gene Therapies (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATX-MTM-002; 2024-512637-32 (Other: CTIS (EU))
Record Dates: First submitted 2017-06-21; First posted 2017-06-27 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: X-Linked Myotubular Myopathy
Keywords: AAV8-Delivered Gene Therapy; XLMTM; Adeno Associated Virus
MeSH Terms: conditions — Myopathies, Structural, Congenital

STUDY DESIGN:
Intervention Model Description: ASPIRO was being conducted in two parts. Part 1 was a dose escalation phase that was evaluating the preliminary safety and efficacy of resamirigene bilparvovec at doses of 1.3x10^14 vg/kg and 3.5x10^14 vg/kg. Part 2 of ASPIRO was a pivotal expansion cohort designed to confirm the safety and efficacy of resamirigene bilparvovec at a dose of 3.5x10^14 vg/kg. The pivotal expansion cohort enrolled eight subjects, consisting of four age-matched pairs (within +/- 6 months of age). One subject from each pair was randomized to receive a single dose of resamirigene bilparvovec at 3.5x10^14 vg/kg, and the other served as a delayed treatment control. Eligible delayed treatment control subjects administered resamirigene bilparvovec after that individual subject completed the Week 24 visit as a delayed treatment control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1.3 × 10^14 vg/kg (Low dose) (Experimental): Participants received 1.3 x 10^14 viral genomes per kilogram (vg/kg) of body weight resamirigene bilparvovec as a single dose intravenously on Day 1. A sentinel dose was given to first participant and if there were no safety concerns, subsequent participants received either resamirigene bilparvovec at the same dose or control with delayed treatment after at least 4 weeks of post-dose data from the sentinel participant.
  Interventions: Genetic: Resamirigene bilparvovec
- 3.5 × 10^14 vg/kg (High dose) (Experimental): Participants received 3.5 × 10^14 vg/kg of body weight resamirigene bilparvovec as a single dose intravenously on Day 1. A sentinel dose was given to first participant and if there were no safety concerns, subsequent participants received either resamirigene bilparvovec at the same dose or control with delayed treatment after at least 4 weeks of post-dose data from the sentinel participant.
  Interventions: Genetic: Resamirigene bilparvovec

INTERVENTIONS:
Genetic: Resamirigene bilparvovec — Resamirigene bilparvovec is an AAV8 vector containing a functional copy of the human MTM1 (hMTM1) gene.
  Other Names: AT132

SUMMARY:
X-linked myotubular myopathy (XLMTM) is a rare and serious condition present at birth where the muscles do not work properly. There are currently no therapies for this serious condition.

The protein myotubularin is needed for muscle development and movement. A gene called MTM1 tells the body to make myotubularin. XLMTM is caused by changes, or mutations, in the MTM1 gene. Changes in the MTM1 gene causes low levels of myotubularin to be made, so the muscles do not work properly. XLMTM may also affect the liver, and in some cases, this can be dangerous and threaten the patient´s life.

Gene therapy is a way of getting a healthy copy of a gene into the body. This allows the body's cells to make a normal protein that may reduce disease symptoms. AT132 is a gene therapy that gets a healthy MTM1 gene into the body to help improve muscle development and function in young children with the disease. AT132 does not treat liver disease, and because of the way the treatment works, it may make liver problems worse.

AT132 was the gene therapy treatment given to children who participated in this study and is not available to the public. In this study, AT132 was given to children for the first time. Due to the occurrence of severe complications and fatalities associated with administration of AT132, the study has been stopped and no further participants will be enrolled.

The main aim of the study is to check how long young children need machines to support breathing (ventilation support) after AT132.

Due to the occurrence of severe complications and fatalities associated with administration of AT132, the study has been stopped and no further participants will be enrolled. This study included children with XLMTM under 5 years old who had breathing problems caused by XLMTM. They couldn't take part if they were born prematurely, recently had surgery, had liver disease or other condition or disease the study doctor thought was medically important. The study did enroll participants with medically significant liver disease.

This is an open-label study. This means that young children and their caregivers, and clinic staff know that young children received AT132. This study was designed with 2 parts and is now in a long-term follow-up phase to collect information on the safety and improvements in muscle function in the children who received AT132.

In Part 1, small groups of young children were given different doses of AT132, with one group receiving a lower dose and one group receiving a higher dose of AT132. The purpose of giving the two doses was to determine which dose was best for treating the muscle disease. After receiving AT132, a medical panel of experts reviewed each child for safety and for how their muscles responded. AT132 did not demonstrate appropriate safety at either dose. Administration of AT132 was stopped. Children who received AT132 are being monitored for 10 years for safety and to understand how their muscles function over time.

DETAILED DESCRIPTION:
This study evaluated safety and efficacy of gene transfer in X-Linked Myotubular Myopathy. Participants received a single dose of resamirigene bilparvovec delivered intravenously.

ASPIRO was being conducted in two parts. Part 1 was a dose escalation phase that was evaluating the preliminary safety and efficacy of Resamirigene bilparvovec at doses of 1.3x10^14 vg/kg and 3.5x10^14 vg/kg. Part 2 of ASPIRO was a pivotal expansion cohort designed to confirm the safety and efficacy of resamirigene bilparvovec at a dose of 3.5x10^14 vg/kg. The pivotal expansion cohort enrolled eight participants, consisting of four age-matched pairs (within +/- 6 months of age). One participant from each pair was randomized to receive a single dose of resamirigene bilparvovec at 3.5x10^14 vg/kg, and the other served as a delayed treatment control. Eligible delayed treatment control participants administered resamirigene bilparvovec after that individual participant completed the Week 24 visit as a delayed treatment control.

The primary efficacy endpoint measures assessed at Week 24. Participants were followed for a total of 10 years after administration of resamirigene bilparvovec. Only Part 1 of the study was reported.

This study utilized an independent Data Monitoring Committee (DMC) that monitored participant safety and provided recommendations to Astellas regarding dose escalation, dose expansion, and safety matters.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of XLMTM resulting from a genetically confirmed mutation in the MTM1 gene as assessed by a Sponsor-approved testing facility.
* Subject is male.
* Subject is aged less than 5 years old at dosing
* Subject requires mechanical ventilatory support:

Part 1: Subject requires some mechanical ventilatory support (e.g., ranging from 24 hours per day full time mechanical ventilation, to noninvasive support such as continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP) during sleeping hours).

Part 2: Subject requires invasive mechanical ventilatory support ranging from 20 - 24 hours per day at screening (confirmed by daytime polysomnographic study).

* Subject requiring invasive mechanical ventilator support is fitted with or willing to be fitted with a cuffed tracheostomy tube for some respiratory assessments.
* Subject has ventilator maximum positive end-expiratory pressure (PEEP) <8 cm H2O at screening.
* UNIQUE to France: Subject's weight is ≥ 4.8 kg.

Exclusion Criteria:

* Subject is participating in an interventional study designed to treat XLMTM.
* Subject born <35 weeks gestation who is still not term as per corrected age.
* Subject tests positive for AAV8 neutralizing antibody with titers above protocol specified threshold.
* Subject had recent surgery (<3 months before Day 1) or has planned surgery that may confound data collection during the first 48 weeks of the study.
* Subject has a clinically important condition other than XLMTM in the opinion of the investigator.
* Subject has a clinically significant underlying liver disease.
* Subject is currently experiencing a clinically important respiratory infection or other active infection.
* Subject has received pyridostigmine or any medication to treat XLMTM within 3 months before Day 1.
* Other than as required per protocol, subject has received immune-modulating agents within 3 months before Day 1 (use of inhaled corticosteroids to manage chronic respiratory conditions is allowed); use of other concomitant medications to manage chronic conditions must have been stable for at least 4 weeks before dosing.
* Subject has a contraindication to prednisolone.
* Subject has a contraindication to study drug or ingredients.
* Subject has previous scoliosis repair surgery/procedure, or planned/expected scoliosis repair surgery/procedure in the 12 months following Day 1 (Part 2 including any subjects enrolled under protocol v8 and beyond).
* Subject has contractures, scoliosis, or other medical condition that would limit the potential to achieve unassisted sitting, in the opinion of the investigator (Part 2 including any subjects enrolled under protocol V8 and beyond).
* Subject is able to sit without assistance for at least 30 seconds at screening, in the opinion of the investigator (Part 2 including any subjects enrolled under protocol V8 and beyond).
* Subject has a clinically important condition, including CTCAE v4.03 Grade ≥ 2 anemia (< 10 g/dL hemoglobin).
* Subject has a contraindication to ursodiol (ursodeoxycholic acid).
* UNIQUE to France: Subject has a prior diagnosis or history of cardiac arrhythmias, myocarditis, or any other cardiac disease.
* UNIQUE to France: Subject has a contraindication to general anesthesia and to muscle biopsy procedures.

Max Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2030-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (6):
- United States (3):
  - UCLA Medical Center, Los Angeles, California
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - National Institute of Neurological Disorders and Stroke/NIH Porter, Bethesda, Maryland
- Hospital for Sick Children, Toronto, Ontario, Canada
- Hopital Armad Trousseau, Paris, France
- Kinderklinik und Kinderpoliklinik im Dr. Von Haunerschen Kinderspital Klinikum der Universitat Munchen, München, Germany

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Shieh PB, Kuntz NL, Dowling JJ, Muller-Felber W, Bonnemann CG, Seferian AM, Servais L, Smith BK, Muntoni F, Blaschek A, Foley AR, Saade DN, Neuhaus S, Alfano LN, Beggs AH, Buj-Bello A, Childers MK, Duong T, Graham RJ, Jain M, Coats J, MacBean V, James ES, Lee J, Mavilio F, Miller W, Varfaj F, Murtagh M, Han C, Noursalehi M, Lawlor MW, Prasad S, Rico S. Safety and efficacy of gene replacement therapy for X-linked myotubular myopathy (ASPIRO): a multinational, open-label, dose-escalation trial. Lancet Neurol. 2023 Dec;22(12):1125-1139. doi: 10.1016/S1474-4422(23)00313-7. PMID 37977713
- See also: Related Info — https://doi.org/10.1016/S1474-4422(23)00313-7

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with X-linked myotubular myopathy (XLMTM) resulting from a genetically confirmed mutation in the myotubular myopathy (MTM) 1 gene as assessed by a Sponsor-approved testing facility were enrolled in this study.
Pre-assignment Details: Participants who met all inclusion criteria and none of the exclusion criteria were enrolled in the study. The study is ongoing, and data for efficacy is reported for Part 1 (week 24) of the study only with mortality and safety data being reported up to data cut-off date 30 June 2023 (up to 5 years).
Groups:
- 1.3 × 10^14 vg/kg (Low Dose): Participants received 1.3 x 10^14 vg/kg of body weight resamirigene bilparvovec as a single dose intravenously on Day 1. A sentinel dose was given to first participant and if there were no safety concerns, subsequent participants received either resamirigene bilparvovec at the same dose or control with delayed treatment after at least 4 weeks of post-dose data from the sentinel participant.
Period: Overall Study
Arm/Group | 1.3 × 10^14 vg/kg (Low Dose) | 3.5 × 10^14 vg/kg (High Dose)
Started | 7 | 20
Delayed Treatment Control (DTC) Group | 1 | 6 (2 participants were randomized but did not receive study intervention.)
Immediate Treatment Group | 6 | 14 (1 participant was randomized but did not receive study intervention.)
Completed | 0 | 0
Not Completed | 7 | 20
Not completed — Randomized, not treated | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 3
Not completed — Ongoing | 5 | 14

BASELINE CHARACTERISTICS:
Population: Included all participants who were randomized in the study.
Groups:
- 1.3 x 10^14 vg/kg (Low Dose): Participants received 1.3 x 10^14 vg/kg of body weight resamirigene bilparvovec as a single dose intravenously on Day 1. A sentinel dose was given to first participant and if there were no safety concerns, subsequent participants received either resamirigene bilparvovec at the same dose or control with delayed treatment after at least 4 weeks of post-dose data from the sentinel participant.
- 3.5 x 10^14 vg/kg (High Dose): Participants received 3.5 × 10^14 vg/kg of body weight resamirigene bilparvovec as a single dose intravenously on Day 1. A sentinel dose was given to first participant and if there were no safety concerns, subsequent participants received either resamirigene bilparvovec at the same dose or control with delayed treatment after at least 4 weeks of post-dose data from the sentinel participant.
- Total: Total of all reporting groups
Arm/Group | 1.3 x 10^14 vg/kg (Low Dose) | 3.5 x 10^14 vg/kg (High Dose) | Total
Number analyzed (Participants) | 7 | 20 | 27
Age, Continuous [Mean (Standard Deviation); unit: Months] | 21.78 (15.47) | 37.66 (24.55) | 33.54 (23.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 20 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 4 | 13 | 17
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 7 | 14 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Ventilation Support [Mean (Standard Deviation); unit: hours] — The hours of ventilation support was based on diary data from participants for whom diary data was collected at baseline and by assessment of time off ventilator questionnaire for all other participants. Baseline is defined as the average of the diary data values in the 7 days leading up to and including the day of administration of the study drug (i.e. Analysis Day - 6 through Day 1). Population: Full Analysis Set (FAS) population (included all randomized and enrolled participants who received resamirigene bilparvovec and had at least 1 post-dose efficacy assessment) with available data was reported.
  hours
    number analyzed (Participants) | 7 | 16 | 23
    (all) | 21 (4.69) | 23.71 (0.52) | 22.89 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hours of Ventilation Support at Week 24
Description: The hours of ventilation support were based on diary data from participants for whom diary data was collected at baseline and by assessment of time off ventilator questionnaire for all other participants. Weekly scores were the average of ventilation hours needed for at least 5 out of the 7 days leading up to and including the analysis visit day (e.g., Day 168 for Week 24). For cases where the diary or the ventilator assessment indicated the ventilator type = "None", then zero was imputed for the number of hours on ventilator.
Time Frame: Baseline, week 24
Population: FAS population. Participants with available data were reported.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1.3 × 10^14 vg/kg (Low Dose) | 3.5 × 10^14 vg/kg (High Dose)
Number analyzed (Participants) | 6 | 16
hours | -8.92 (9.31) | -5.84 (5.45)

2. Secondary Outcome: Percentage of Participants Achieving Functionally Independent Sitting for At Least 30 Seconds by Week 24
Description: Independence to sit is defined as a participant who sits for at least 30 seconds without assistance from another person or object. Data was determined from the motor milestone electronic case report form (eCRF) or the Bayley Scales of Infant and Toddler Development (BSID) subtest performance criteria number 26, used to determine whether the participant achieves (Yes) or doesn't achieve (No) the milestone. If data was not available then they would be included as "missing".
Time Frame: Week 24
Population: FAS population. Participants with available data were reported.
Measure: Number; unit: Percentage of participants
Arm/Group | 1.3 × 10^14 vg/kg (Low Dose) | 3.5 × 10^14 vg/kg (High Dose)
Number analyzed (Participants) | 6 | 13
Percentage of participants
  Achieved | 83.3 | 61.5
  Not Achieved | 16.7 | 38.5

3. Secondary Outcome: Time to Reduction in Required Ventilator Support to ≤ 16 Hours a Day From Dosing to Week 24
Description: The reduced ventilator time was obtained directly from the daily diary or assessment of the time off ventilator questionnaire. The first instance of time reduction reported as ≤ 16 hours per day was considered as an event. Kaplan- Meier estimate was used for analysis.
Time Frame: Baseline up to week 24
Population: FAS population. Participants with available data were reported.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | 1.3 × 10^14 vg/kg (Low Dose) | 3.5 × 10^14 vg/kg (High Dose)
Number analyzed (Participants) | 6 | 17
Weeks | 12.1 [4.1 to 16.1] | NA [17.1 to NA] — Data was not estimable because less than 50% of participants had event (data was estimated using Kaplan-Meier [KM] and it requires at least 50% of event to be able to calculate time using KM).

4. Secondary Outcome: Change From Baseline in Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) Total Score at Week 24
Description: The CHOP INTEND is an assessment scale that was originally designed to quantify motor abilities in infants aged 1.4 to 37.9 months, with spinal muscular atrophy type I (SMA-I) and has been validated for X-linked myotubular myopathy (XLMTM). The scale contains 16 questions, each of which is scored on a scale of 0 to 4, with 0 being no response/ability to perform the movement and 4 highest abilities to perform the task, per CHOP INTEND item instructions. The score used for analysis is the total sum of all 16 questions, which will range from 0 to 64. Higher score indicates better neuromuscular function. If an item is missing or scored as "Could Not Test (CNT)" then 0 will be imputed for the item score.
Time Frame: Baseline, week 24
Population: FAS population. Participants with available data were reported.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | 1.3 × 10^14 vg/kg (Low Dose) | 3.5 × 10^14 vg/kg (High Dose)
Number analyzed (Participants) | 7 | 12
Score on scale | 11.86 (15.12) | 13.25 (13.35)

5. Secondary Outcome: Change From Baseline in Maximal Inspiratory Pressure (MIP) at Week 24
Description: MIP is a quick and non-invasive test to measure strength of inspiratory muscles, primarily diaphragm, and allows for assessment of ventilatory failure, restrictive lung disease and respiratory muscle strength. MIP refers to how much air pressure force an individual creates by inhaling through the mouth as hard as possible.
Time Frame: Baseline, week 24
Population: FAS population. Participants with available data were reported.
Measure: Mean (Standard Deviation); unit: centimeter of water (cmH2O)
Arm/Group | 1.3 × 10^14 vg/kg (Low Dose) | 3.5 × 10^14 vg/kg (High Dose)
Number analyzed (Participants) | 7 | 12
centimeter of water (cmH2O) | 41.07 (35.03) | 26.72 (28.35)

6. Secondary Outcome: Change From Baseline in Quantitative Analysis of Myotubularin Expression in the Muscle Biopsy at Week 24
Description: Myotubularin is a protein, a highly conserved, dual-specific lipid phosphatase that is involved in the development, maturation, and maintenance of skeletal muscle cells. Myotubularin is encoded by an MTM1 gene. The concentration of the sample was normalized such that the equivalent amount of protein was tested per sample.
Time Frame: Baseline, week 24
Population: FAS population. Participants with available data were reported.
Measure: Mean (Standard Deviation); unit: picograms (pg)/15 microgram(µg) protein
Arm/Group | 1.3 × 10^14 vg/kg (Low Dose) | 3.5 × 10^14 vg/kg (High Dose)
Number analyzed (Participants) | 7 | 10
picograms (pg)/15 microgram(µg) protein | 923.69 (816.09) | 2848.40 (2903.83)

7. Secondary Outcome: Change From Baseline in Quality of Life Assessment of Caregiver Experience With Neuromuscular Disease (ACEND) Total Score at Week 24
Description: ACEND was developed to measure impact on lives of parents/legally authorized representatives /caregivers caring for children with severe neuromuscular disorders. ACEND has 41 items which reflected 2 domains (physical impact [feeding/grooming/dressing {6 items}, sitting/play {5 items}, transfers {5 items} and mobility {7 items}] and general caregiver impact [time {4 items}, emotion {9 items}, and finance {5 items}]). Score for each item was based on 6- or 5-point ordinal scale, and scores for each domain and subdomain were scored on 0 - 100 scale. Higher scores reflected caregivers experiencing less intense care-giving impact. Raw scores for each subdomain was created by computing algebraic mean of items for those respondents who completed one item or more; setting missing for those items with no responses. Then, arithmetic mean of responded items was standardized to 0 to 100 score and transformed scores were from 0 to 100 for each subdomain. Higher score indicated a better outcome.
Time Frame: Baseline, week 24
Population: FAS population. Participants with available data were reported.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | 1.3 × 10^14 vg/kg (Low Dose) | 3.5 × 10^14 vg/kg (High Dose)
Number analyzed (Participants) | 7 | 15
Score on scale | 20.12 (18.81) | 13.82 (12.33)

8. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Inventory (PedsQL) Assessment Total Score at Week 24
Description: PedsQL is a tool designed to measure health-related quality of life in healthy children and adolescents and those with acute and chronic health conditions. PedsQL measures the core dimensions of health as delineated by the World Health Organization, as well as role (school) functioning. This questionnaire has different modules that are administered depending on the age and condition of the child. Each item of the questionnaire is measured on a 5-point likert scale from - 0 (Never) to 4 (Almost always). The module is composed of 25 items comprising 3 dimensions: About My Neuromuscular Disease (17 items), Communication (3 items), About Our Family Resources (5 items). Items are reversed scored and linearly transformed to a total score of 0-100 scale. Higher scales/scores indicate lower problems.
Time Frame: Baseline, week 24
Population: FAS population. Participants with available data were reported.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | 1.3 × 10^14 vg/kg (Low Dose) | 3.5 × 10^14 vg/kg (High Dose)
Number analyzed (Participants) | 7 | 15
Score on scale | 9.39 (15.51) | 12.06 (19.23)

9. Secondary Outcome: Mean Percent of Age-appropriate Clinically Relevant Gross Motor Function Milestones Attained Through Week 24
Description: Motor Developmental Milestones included: head control (holds head erect for at least 15 seconds without support), rolls from back to sides (turns from back to both sides), sits without support (sits alone without support for at least 10 seconds), stands with assistance (supports own weight for at least 2 seconds), crawls (makes forward progress of at least 5 feet by crawling on hands and knees), pulls to stand (raises self to standing position using chair or other convenient object for support), walks with assistance (child walks by making coordinated, alternating stepping movements. May hold on with 1 or 2 hands for support), stands alone (stands alone for at least 3 seconds after you release hands), walks alone (takes at least 3 steps without support, even if gait is stiff-legged and wobbly). Mean percentage of gross motor function milestones attained was reported.
Time Frame: Baseline, weeks 4, 12, 16 and 24
Population: FAS population. Participants with available data were reported.
Measure: Mean (Standard Deviation); unit: Percentage of gross motor function
Arm/Group | 1.3 × 10^14 vg/kg (Low Dose) | 3.5 × 10^14 vg/kg (High Dose)
Number analyzed (Participants) | 2 | 10
Percentage of gross motor function
  Baseline: number analyzed (Participants) | 1 | 8
  Baseline | 0.0 | 12.50 (15.81)
  Week 4: number analyzed (Participants) | 2 | 6
  Week 4 | 30.00 (28.28) | 23.33 (19.66)
  Week 12: number analyzed (Participants) | 1 | 9
  Week 12 | 0.0 | 26.85 (15.06)
  Week 16: number analyzed (Participants) | 1 | 10
  Week 16 | 0.0 | 25.25 (16.26)
  Week 24: number analyzed (Participants) | 1 | 9
  Week 24 | 0.0 | 26.67 (19.36)

10. Secondary Outcome: Percentage of Participants Achieving Full Ventilator Independence at Week 24
Description: "Full ventilator independence" is defined as: the date of removal from ventilator field on the "Assessment of Ventilator Parameters" eCRF is not blank or "Is subject on a ventilator" = "No" on the same eCRF.
Time Frame: Week 24
Population: FAS population. Participants with available data were reported.
Measure: Number; unit: Percentage of participants
Arm/Group | 1.3 × 10^14 vg/kg (Low Dose) | 3.5 × 10^14 vg/kg (High Dose)
Number analyzed (Participants) | 7 | 16
Percentage of participants
  Achieved | 28.6 | 0
  Not Achieved | 71.4 | 100

11. Secondary Outcome: Duration of Overall Survival
Description: Survival status was assessed at each visit until the participant withdraws consent or completes the study. If the participant missed a visit or withdraws for a reason other than withdrawal of consent or death, the site contacted the parent(s)/legally authorized representatives to ascertain if the participant was alive. For participants who withdrew from the study, the participant was contacted every 6 months for 5 years after administration and to assess for survival. Kaplan- Meier estimate was used for analysis.
Time Frame: Baseline up to 5 years
Population: FAS population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1.3 × 10^14 vg/kg (Low Dose) | 3.5 × 10^14 vg/kg (High Dose)
Number analyzed (Participants) | 7 | 17
Months | NA [2.10 to NA] — Data was not estimable because less than 50% of participants had event (data was estimated using KM and it requires at least 50% of event to be able to calculate time using KM). | NA [NA to NA] — Data was not estimable because less than 50% of participants had event (data was estimated using KM and it requires at least 50% of event to be able to calculate time using KM).

12. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a participant administered a study drug not necessarily having a causal relationship with this treatment. An AE can therefore be any unfavorable & unintended sign, symptom, or disease temporally associated with the use of medicinal product (MP) whether or not considered related to MP. A TEAE is any AEs, regardless of relationship to study drug, that begins or worsens on or after baseline (dosing) visit date.
Time Frame: From first dose to 5 years
Population: Safety Analysis Set (SAF) consisted of all randomized participants who received resamirigene bilparvovec.
Measure: Number; unit: Participants
Arm/Group | 1.3 × 10^14 vg/kg (Low Dose) | 3.5 × 10^14 vg/kg (High Dose)
Number analyzed (Participants) | 7 | 17
Participants | 7 | 17

ADVERSE EVENTS:
Time Frame: From first dose to 5 years
Description: All-cause mortality and AEs included SAF population that consisted of all randomized participants who received resamirigene bilparvovec.
Arm/Group | 1.3 x 10^14 vg/kg (Low Dose) | 3.5 x 10^14 vg/kg (High Dose)
All-Cause Mortality (participants affected / at risk) | 1/7 | 3/17
Serious Adverse Events (participants affected / at risk) | 5/7 | 13/17
Other Adverse Events (participants affected / at risk) | 7/7 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.3 x 10^14 vg/kg (Low Dose) (N=7) | 3.5 x 10^14 vg/kg (High Dose) (N=17)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Combined immunodeficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 3 (4)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Protein-losing gastroenteropathy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 2 (5)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Immune system disorder (Immune system disorders) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (2)
Septic shock (Infections and infestations) | 1 (2) | 0 (0)
Serratia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (2) | 2 (5)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Troponin I increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epiglottic oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Withdrawal hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.3 x 10^14 vg/kg (Low Dose) (N=7) | 3.5 x 10^14 vg/kg (High Dose) (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (4)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 9 (11)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Coronary sinus dilatation (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 2 (2) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Dolichocephaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Laryngeal cleft (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Portal venous system anomaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Talipes (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Precocious puberty (Endocrine disorders) | 1 (1) | 1 (1)
Astigmatism (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 6 (9)
Diarrhoea (Gastrointestinal disorders) | 3 (8) | 3 (7)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 1 (1)
Teething (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (3) | 9 (13)
Catheter site extravasation (General disorders) | 0 (0) | 1 (1)
Developmental delay (General disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Medical device site granuloma (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (3)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (9) | 10 (14)
Secretion discharge (General disorders) | 0 (0) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 6 (6)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 2 (3)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (4) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic oedema (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial tracheitis (Infections and infestations) | 2 (2) | 2 (6)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2) | 4 (4)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Coxsackie viral infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 2 (2)
Ear infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Enterobiasis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal bacterial overgrowth (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2) | 2 (4)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (2) | 0 (0)
Otitis media (Infections and infestations) | 4 (7) | 4 (5)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Otitis media staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (2) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 3 (4)
Respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (2)
Rhinovirus infection (Infections and infestations) | 1 (1) | 1 (2)
Scarlet fever (Infections and infestations) | 0 (0) | 2 (2)
Skin candida (Infections and infestations) | 0 (0) | 2 (2)
Tracheitis (Infections and infestations) | 0 (0) | 1 (4)
Tracheostomy infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (6) | 7 (15)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 4 (9) | 5 (7)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 4 (5)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma site hypergranulation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 1 (2) | 3 (3)
Aldolase increased (Investigations) | 0 (0) | 1 (1)
Ammonia increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 4 (4)
Bile acids increased (Investigations) | 2 (2) | 2 (3)
Bilirubin urine (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase decreased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase BB increased (Investigations) | 1 (1) | 1 (1)
Blood creatine phosphokinase MB increased (Investigations) | 1 (1) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 5 (9) | 6 (7)
Blood fibrinogen decreased (Investigations) | 0 (0) | 1 (1)
Blood immunoglobulin G decreased (Investigations) | 0 (0) | 1 (1)
Blood iron increased (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 2 (2)
Blood osmolarity increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1)
Blood zinc decreased (Investigations) | 0 (0) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 3 (3) | 5 (6)
Carbon dioxide decreased (Investigations) | 0 (0) | 1 (1)
Cardiac imaging procedure abnormal (Investigations) | 0 (0) | 1 (1)
Complement factor decreased (Investigations) | 1 (1) | 0 (0)
Cytokine increased (Investigations) | 1 (1) | 0 (0)
Echocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Electrocardiogram ST segment elevation (Investigations) | 0 (0) | 1 (1)
Electrocardiogram low voltage (Investigations) | 0 (0) | 1 (1)
Faecal fat increased (Investigations) | 0 (0) | 1 (1)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (3) | 3 (3)
Haptoglobin decreased (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (2)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Human rhinovirus test positive (Investigations) | 0 (0) | 1 (1)
Interleukin level increased (Investigations) | 0 (0) | 1 (1)
Interleukin-2 receptor increased (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (2)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte morphology abnormal (Investigations) | 0 (0) | 1 (1)
Myocardial necrosis marker increased (Investigations) | 0 (0) | 1 (1)
Neutrophil toxic granulation present (Investigations) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 1 (2)
Pancreatic enzymes increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Prealbumin decreased (Investigations) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 2 (3) | 0 (0)
Prothrombin time abnormal (Investigations) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 2 (2)
QRS axis abnormal (Investigations) | 1 (1) | 0 (0)
Red blood cell burr cells present (Investigations) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1)
Serum ferritin increased (Investigations) | 0 (0) | 1 (1)
Stool reducing substances increased (Investigations) | 0 (0) | 1 (1)
Thrombin time prolonged (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 3 (3) | 3 (4)
Transferrin decreased (Investigations) | 0 (0) | 1 (1)
Transferrin saturation increased (Investigations) | 0 (0) | 1 (1)
Troponin I increased (Investigations) | 1 (2) | 2 (4)
Troponin T increased (Investigations) | 1 (2) | 5 (6)
Troponin increased (Investigations) | 1 (1) | 2 (2)
Ultrasound liver abnormal (Investigations) | 1 (1) | 0 (0)
Ultrasound scan abnormal (Investigations) | 0 (0) | 1 (1)
Urine sodium decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Feeding intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin A deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Epiphyses delayed fusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Epiphyses premature fusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Extremity contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Language disorder (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (2) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 1 (1) | 2 (2)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Autism spectrum disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Testicular disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular infarction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Epiglottic oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (8)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tracheostomy closure (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT03199469/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT03199469/SAP_001.pdf